CLINICAL TRIAL: NCT06821061
Title: A PHASE 1/2 RANDOMIZED, DOUBLE-BLINDED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND IMMUNOGENICITY OF MODIFIED RNA VACCINE CANDIDATES AGAINST INFLUENZA AND COVID-19 IN HEALTHY INDIVIDUALS
Brief Title: A Study to Learn About How the Flu and COVID-19 Vaccines Act in Healthy People
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C6271001; C6271001-C1 (Other: Alias Study Number); C6271001-C1A (Other: Alias Study Number)
Record Dates: First submitted 2025-02-07; First posted 2025-02-11 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Influenza; COVID-19 (Coronavirus Disease 2019)
MeSH Terms: conditions — Influenza, Human; COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (33):
- Arm A (Experimental): Low Dose COVID-19 Vaccine (1a)
  Interventions: Biological: Investigational COVID-19 Vaccine
- Arm B (Experimental): Low Dose COVID-19 Vaccine ( 1b)
  Interventions: Biological: Investigational COVID-19 Vaccine
- Arm C (Experimental): Low Dose COVID-19 Vaccine ( 1c)
  Interventions: Biological: Investigational COVID-19 Vaccine
- Arm D (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 1)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm E (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (Medium Dose Combination 2)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm F (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 3)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm G (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 4)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm H (Active Comparator): Licensed COVID-19 Vaccine
  Interventions: Biological: Licensed COVID-19 Vaccine
- Arm I (Active Comparator): Licensed Influenza Vaccine (1)
  Interventions: Biological: Licensed Influenza Vaccine 1
- Arm J (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 5)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm K (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 6)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm L (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 7)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm M (Active Comparator): Licensed COVID-19 Vaccine
  Interventions: Biological: Licensed COVID-19 Vaccine
- Arm N (Active Comparator): Licensed Influenza Vaccine (2)
  Interventions: Biological: Licensed Influenza Vaccine 2
- Arm AA (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 6)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm BB (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 4)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm CC (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 7)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm DD (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (Medium Dose Combination 2)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm EE (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 3)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm FF (Active Comparator): Licensed COVID-19 Vaccine
  Interventions: Biological: Licensed COVID-19 Vaccine
- Arm GG (Active Comparator): Licensed Influenza Vaccine (3)
  Interventions: Biological: Licensed Influenza Vaccine 3
- Arm HH (Active Comparator): Licensed Influenza Vaccine (2)
  Interventions: Biological: Licensed Influenza Vaccine 2
- Arm II (Experimental): Low Dose COVID-19 Vaccine ( 1b)
  Interventions: Biological: Investigational COVID-19 Vaccine
- Arm JJ (Experimental): Low Dose COVID-19 Vaccine ( 1c)
  Interventions: Biological: Investigational COVID-19 Vaccine
- Arm KK (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 4)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm LL (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 7)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm MM (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (Medium Dose Combination 2)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm NN (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 3)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm OO (Experimental): Investigational Influenza and COVID-19 Combination Vaccine (High Dose Combination 5)
  Interventions: Combination Product: Investigational Influenza and COVID-19 Combination Vaccine
- Arm PP (Experimental): Medium Dose Investigational Influenza Vaccine (1)
  Interventions: Biological: Investigational Influenza Vaccine
- Arm QQ (Experimental): High Dose Investigational Influenza Vaccine (2)
  Interventions: Biological: Investigational Influenza Vaccine
- Arm RR (Active Comparator): Licensed COVID-19 Vaccine
  Interventions: Biological: Licensed COVID-19 Vaccine
- Arm SS (Active Comparator): Licensed Influenza Vaccine (3)
  Interventions: Biological: Licensed Influenza Vaccine 3

INTERVENTIONS:
Biological: Investigational Influenza Vaccine — Investigational Influenza Vaccine
  Arms: Arm PP; Arm QQ
Biological: Investigational COVID-19 Vaccine — Investigational COVID-19 Vaccine
  Arms: Arm A; Arm B; Arm C; Arm II; Arm JJ
Combination Product: Investigational Influenza and COVID-19 Combination Vaccine — Investigational Combined Influenza and COVID-19 Vaccine
  Arms: Arm AA; Arm BB; Arm CC; Arm D; Arm DD; Arm E; Arm EE; Arm F; Arm G; Arm J; Arm K; Arm KK; Arm L; Arm LL; Arm MM; Arm NN; Arm OO
Biological: Licensed Influenza Vaccine 1 — Licensed Influenza Vaccine 1
  Arms: Arm I
Biological: Licensed Influenza Vaccine 2 — Licensed Influenza Vaccine 2
  Arms: Arm HH; Arm N
Biological: Licensed Influenza Vaccine 3 — Licensed Influenza Vaccine 3
  Arms: Arm GG; Arm SS
Biological: Licensed COVID-19 Vaccine — Pfizer-BioNTech COVID-19 Vaccine
  Arms: Arm FF; Arm H; Arm M; Arm RR

SUMMARY:
The purpose of this study is to learn about how the flu and COVID vaccines act when given alone or when mixed together.

This study is seeking healthy participants aged 18 or older. All participants in this study will receive only 1 shot to their arm, either a flu or COVID vaccine, alone or mixed. Participants will take part in this study for about 6 months, and participants will need to visit the clinical study site at least 4 times.

ELIGIBILITY:
Inclusion criteria:

* Participants 18 years of age or older
* Healthy participants who are determined by medical history, physical examination (if clinically required), and clinical judgement of the investigator to be eligible for inclusion in the study

Exclusion criteria:

* Vaccination with any investigational or licensed influenza vaccine within 150 days of enrollment
* Vaccination with any investigational or licensed COVID 19 vaccine within 150 days of enrollment.
* Receipt of antiviral therapies for influenza (eg, Tamiflu) within 180 days prior to Day 1.

Refer to the study contact for further eligibility details

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2650 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-12-17 (Actual); Study Completion 2025-12-17 (Actual)

PRIMARY OUTCOMES:
Percentage of participants reporting prompted local reactions within 7 days following investigational product administration | Day 7
Percentage of participants reporting prompted systemic events within 7 days following investigational product administration | Day 7
Percentage of participants reporting adverse events (AEs) through 1 month following investigational product administration | 1 month
Percentage of participants reporting serious adverse events (SAEs) through 6 months following investigational product administration | 6 months

SECONDARY OUTCOMES:
GMTs before and through 1 month following investigational product administration | Before vaccination through to 1 month after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (30):
- United States (30):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Orange County Research Center, Lake Forest, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Clinical Research Consulting, Milford, Connecticut
  - Alliance for Multispecialty Research, LLC, Doral, Florida
  - Indago Research & Health Center, Inc, Hialeah, Florida
  - Miami Dade Medical Research Institute, LLC, Miami, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Clinical Research Professionals, Chesterfield, Missouri
  - Las Vegas Clinical Trials, North Las Vegas, Nevada
  - Upstate Global Health Institute, East Syracuse, New York
  - University of Rochester Medical Center, Rochester, New York
  - Trial Management Associates - Wilmington - Floral Parkway, Wilmington, North Carolina
  - Centricity Research Columbus Ohio Multispecialty, Columbus, Ohio
  - DM Clinical Research - Philadelphia, Philadelphia, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - AMR Clinical, Knoxville, Tennessee
  - Clinical Research Associates Inc, Nashville, Tennessee
  - Headlands Horizons, LLC dba Headlands Research-Brownsville, Brownsville, Texas
  - DM Clinical Research- Cyfair, Houston, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Dynamed Clinical Research, LP d/b/a DM Clinical Research, Tomball, Texas
  - J. Lewis Research, Inc. / Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research, Inc. / Foothill Family Clinic South, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Kaiser Permanente Washington Health Research Institute (KPWHRI), Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C6271001